CLINICAL TRIAL: NCT06109987
Title: Clinical Evaluation of High-viscosity Glass-hybrid Systems Compared With a Bulk Fill Composite Resin in Different Cavity Type
Brief Title: Clinical Evaluation of Bulk-fill Restorative Materials
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Muhammet Karadaş, Assistan Professor, Recep Tayyip Erdogan University
Other Study IDs: RTEUDHFMKARADAS002
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-02

CONDITIONS: Caries; Dentin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: World Dental Federation criteria (FDI) — Restorations were evaluated with FDI criteria.

SUMMARY:
High-viscosity glass ionomer cements have been developed to improve the weak mechanical properties of glass ionomer cements, increase wear resistance and improve their limited indications. There are limited clinical studies on the use of high-viscosity glass ionomer cements in areas with large cavities bearing stress. The aim of this study is to compare the clinical performance of two different high-viscosity glass ionomer cements with a bulk-fill resin composite in different cavities.

DETAILED DESCRIPTION:
This study was a double-blind (evaluator and patient) randomized controlled clinical study with three study groups with an equal allocation. Three different restorative materials were compared in Class I, II, and V restorations.

The treated patients were called back for controls after one week, six months, and eighteen months. Restorations were evaluated clinically according to modified FDI criteria. In terms of marginal discoloration, fracture and retention, marginal adaptation, post-operative sensitivity, secondary caries, color match and difference criteria were examined.

Clinical evaluation was performed by one qualified clinicians using a mirror and probe under reflector light. Bite-wing radiographs were taken from the patients who were called for controls at 6-moth and 18-month to evaluate the formation of secondary caries.

Differences between adhesives at each time period were evaluated using Fisher's Exact test. The effect of time on restorations was evaluated using Wilcoxon Signed rank test (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreed to participate in the study after being informed about the study.
* Volunteer must not be under 18 years of age
* No systemic disease
* Having healthy oral hygiene
* As a result of clinical and radiographic examination, there is a carious lesion at D1 and D2 levels according to the caries classification method.
* The tooth to be restored is vital

Exclusion Criteria:

* Refusal to participate in the study after being informed about the study
* The patient has a history of teeth grinding
* Volunteer must be under 18 years of age
* The volunteer is undergoing or will begin orthodontic treatment
* The volunteer has a serious systemic disease
* The tooth to be restored has endodontic and periodontal problems
* Volunteer's pregnancy status
* Extraction of one of the teeth opposite or in contact with the tooth to be restored

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Teeth with primary caries that extends into the middle or outer one-third of the dentin (D1 or D2) in radiographs were included in the study. Visually, teeth with visible signs of enamel breakdown or moderate demineralization of dentin (ICDAS 4) in occlusal and smooth surfaces were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-09-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of different restorative materials | Baseline
  Restored teeth were evaluated according to FDI criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet 53 Karadaş, PhD, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Muhammet Karadaş, Rize, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT06109987/Prot_000.pdf